CLINICAL TRIAL: NCT07017283
Title: Effect of Deep Analgosedation vs. Endotracheal Intubation General Anesthesia on Perioperative Respiratory Adverse Events in Elderly ERCP Patients: An Open-Label Randomized Controlled Trial
Brief Title: Effect of Deep Analgosedation vs. Endotracheal Intubation General Anesthesia on on Perioperative Sedation Related Adverse Events in Elderly ERCP Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gang Chen (Other)
Responsible Party: Sponsor-Investigator, Gang Chen, chief physician, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERCP
Record Dates: First submitted 2025-05-21; First posted 2025-06-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Biliary and Pancreatic Diseases; Endoscopic Retrograde Cholangiopancreatography (ERCP)
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator)
  Interventions: Device: Tracheal intubation general anesthesia
- Deep sedation (Experimental)
  Interventions: Device: Nasopharyngeal airway ventilation

INTERVENTIONS:
Device: Tracheal intubation general anesthesia — Endotracheal intubation with general anesthesia was administered to the patient during the ERCP procedure.
  Arms: General anesthesia
Device: Nasopharyngeal airway ventilation — Nasopharyngeal airway-assisted deep sedation was employed for the patient during the ERCP procedure.
  Arms: Deep sedation

SUMMARY:
This study aims to investigate the impact of deep analgosedation versus endotracheal intubation general anesthesia on perioperative sedation related adverse events in elderly ERCP patients.

DETAILED DESCRIPTION:
This study aims to investigate the impact of deep analgosedation versus endotracheal intubation general anesthesia on perioperative sedation related adverse events in elderly ERCP patients.

ELIGIBILITY:
Inclusion criteria：

1. Aged 60 and above;
2. ASA physical status≤III;
3. Patients who scheduled for elective therapeutic ERCP (ERCP complexity grading system;
4. Willing to provide informed consent (or by legal guardian/witness if applicable).

Exclusion criteria：

1: Altered gastrointestinal anatomy, delayed gastric emptying, or gastric outlet obstruction； 2.Coagulopathy or epistaxis tendency; 3.Cardiac diseases (e.g., coronary artery disease, heart failure, arrhythmias); 4.Pulmonary diseases (e.g., asthma, COPD); 5.Prior hypersensitivity to anesthetic agents; 6.Active upper respiratory infection； 7.Severe liver and kidney diseases； 8.Difficult airway: Preoperative anesthesiologist assessment of difficult airway； 9.Psychiatric disorders, cognitive impairment, critical illness, or pregnancy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Perioperative sedation related adverse events | Perioperative period

SECONDARY OUTCOMES:
recovery room time | Perioperative period
Nasopharyngeal airway requires face mask ventilation or switching to tracheal intubation | Perioperative
Second intubation after the tracheal intubation is removed | Perioperative
Tachycardia (>100 beats/minute) or bradycardia (<50 beats/minute) | Perioperative
Rating of reflux degree | perioperative
QoR-15 score on POD1 | Postoperative day 1
Incidence of postoperative nausea and vomiting | postoperative day 1
respiratory failure/ARDS incidence | Perioperative
Postoperative cognitive function assessment (MoCA) | Perioperative
  The Montreal Cognitive Assessment (MoCA) has a total score of 30 points, with a score of ≥26 considered normal
patient/endoscopist satisfaction | Perioperative
  Patient/endoscopist satisfaction with sedation type was assessed using a 10-point visual analog scale (VAS), where 1 represented the worst possible experience and 10 indicated the optimal experience
hospital stay duration | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhijiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol